CLINICAL TRIAL: NCT01155050
Title: Louisiana State University Health Care Services Division (LSUHCSD) Tele-Health Projects: Weight Loss in Chronic Disease Patient Population
Brief Title: Weight Loss in Chronic Disease Patient Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PBRC 29032
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Results first posted 2020-12-29 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Overweight; Obesity; Diabetes; Hypertension
Keywords: overweight; obese; type II diabetes; hypertension
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus; Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The study randomized consenting subjects to four arms for evaluation of different weight loss strategies.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tele-health Home Monitoring (Active Comparator): Participants will use the tele-health monitoring equipment to measure daily weight.
  Interventions: Device: Tele-health Home Monitoring
- Self-Directed Group (No Intervention): Participants will receive information on physical activity recommendations and guidelines on nutrition aimed at promoting weight loss.
- TrestleTree Telephone Coaching (Active Comparator): Participants will speak to Trestletree health coaches for 15 to 60 minutes each session. During these sessions, the coaches will identify the participant's stage of change and intervene accordingly. The telephone calls will be centered on weight loss.
  Interventions: Behavioral: TrestleTree Telephone Coaching
- Home monitoring + telephone coach (Active Comparator): System to track stage of change in weight loss.
  Interventions: Device: Tele-health Home Monitoring Plus Trestle Telephone Coaching

INTERVENTIONS:
Device: Tele-health Home Monitoring — Daily tele-health monitoring data will be collected from randomized participants.
  Other Names: Home Monitoring
  Arms: Tele-health Home Monitoring
Behavioral: TrestleTree Telephone Coaching — Weekly or bi-weekly phone calls from TrestleTree health coaches with a focus on weight loss.
  Other Names: Telephone Coaching
  Arms: TrestleTree Telephone Coaching
Device: Tele-health Home Monitoring Plus Trestle Telephone Coaching — Daily collection of data through the tele-health home monitor and weekly or bi-weekly phone calls with a Trestletree Health Coach.
  Other Names: Home Monitoring and telephone coaching
  Arms: Home monitoring + telephone coach

SUMMARY:
This study will assess the effect of in-home tele-health monitoring on health outcomes for LSUHCSD chronic disease, overweight or obese patients diagnosed with type II diabetes or hypertension.

DETAILED DESCRIPTION:
This study will assess the effect of in-home tele-health monitoring on health outcomes for LSUHCSD chronic disease, overweight or obese patients diagnosed with type II diabetes or hypertension. Primary emphasis will be on assessing the effect of tele-health home monitoring combined with motivational telephone coaching on weight loss and waist circumference as compared to self-directed, home monitoring alone, and telephone coaching alone. Secondary outcomes such as blood pressure, Hemoglobin A1c (HbA1c), fasting blood sugar, and cholesterol will be examined as well.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 yrs old
* BMI ≥ 25 kg/m2 and waist circumference > 40 inches (men)/ 35 inches (women)
* Weight ≤ 500lbs
* At least one of the following:
* Fasting blood sugar > 100 mg/dL at any point and/or taking medications for diabetes And/Or
* Resting blood pressure > 130/90 mm Hg at any point and/or taking medications for hypertension
* Not involved in regular physical activity or weight loss management programs
* Capable of being physically active
* Physically able to use in-home equipment (or presence of a household member who can assist the subject in equipment use)
* Currently-working conventional telephone line at primary residence
* Grounded electrical power supply at primary residence
* Have been in LSU HCSD system for 6 months and anticipate remaining in the LSU HCSD patient population for the next 6 months

Exclusion Criteria:

* A history of drug abuse in the last year, or excess alcohol consumption (40g/day)6
* Currently dieting or engaging in any activity with the goal of losing weight
* Significant weight loss or weight gain in the past year (> 50 lbs) or current use of weight loss medications
* History of gastrointestinal bypass or other bariatric surgery in the last 3 years
* Diagnosis of congestive heart failure
* Under treatment for end-stage renal disease or end-stage liver disease
* History of major organ transplant
* History of cancers requiring treatment in the past 5 years with anything but excellent prognosis
* Current diagnosis of schizophrenia, bipolar disorder, or other psychotic disorders
* Pregnant or plan on becoming pregnant in the next 12 months.
* Lack support from health care provider or family members.
* Current member of household participating in study
* Factors that may limit adherence to intervention or affect conduct of the trial.
* Unable or unwilling to communicate with staff, to provide written informed consent, or accept the randomized assignment.
* Any other condition, which, in the opinion of the investigators would impede competence or compliance or possibly hinder completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy S. Church, MD, MPH, PhD, Study Chair — Pennington Biomedical Research Center; Donna H. Ryan, MD, Study Chair — Pennington Biomedical Research Center; Valerie H. Myers, PhD, Study Chair — Pennington Biomedical Research Center; Ronald W. Horswell, PhD, Study Chair — Pennington Biomedical Research Center; Monisha Chadha, MD, Principal Investigator — Louisiana State University Health Care Services Division
Locations (3):
- United States (3):
  - Earl K. Long Medical Center, Baton Rouge, Louisiana
  - Leonard J. Chabert Medical Center, Houma, Louisiana
  - WO Moss Regional Medical Center, Lake Charles, Louisiana

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between January 1, 2010 and June 30, 2010. Recruitment was done at primary care clinics at three LSU Health Care Services Division locations in three Louisiana cities.
Pre-assignment Details: Potential subjects were screened for eligibility and then randomized within site to the four treatment arms.
Period: Overall Study
Arm/Group | Tele-health Home Monitoring | Self-Directed Group | TrestleTree Telephone Coaching | Home Monitoring + Telephone Coach
Started | 50 | 51 | 52 | 49
Completed | 35 | 31 | 33 | 27
Not Completed | 15 | 20 | 19 | 22
Not completed — Lost to Follow-up | 15 | 20 | 19 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tele-health Home Monitoring | Self-Directed Group | TrestleTree Telephone Coaching | Home Monitoring + Telephone Coach | Total
Number analyzed (Participants) | 50 | 51 | 52 | 49 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.04 (9.74) | 51.94 (11.73) | 50.62 (9.87) | 49.55 (10.37) | 50.80 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 49 | 48 | 43 | 186
  Male | 4 | 2 | 4 | 6 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 1 | 3 | 9
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 32 | 26 | 28 | 25 | 111
  White | 15 | 23 | 23 | 21 | 82
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 51 | 52 | 49 | 202
Diagnosis of diabetes [Count of Participants; unit: Participants] | 26 | 25 | 23 | 21 | 95
Diagnosis of hypertension [Count of Participants; unit: Participants] | 49 | 47 | 50 | 47 | 193
Use diabetes medication [Count of Participants; unit: Participants] | 24 | 18 | 19 | 21 | 82
Use cholesterol medication [Count of Participants; unit: Participants] | 20 | 30 | 22 | 15 | 87
Use blood pressure medication [Count of Participants; unit: Participants] | 47 | 44 | 47 | 41 | 179
Use anti-depression medication [Count of Participants; unit: Participants] | 12 | 14 | 19 | 15 | 60
Low-density lipoprotein [Mean (Standard Deviation); unit: mg/dL] | 118 (32) | 120 (33) | 117 (41) | 117 (36) | 118 (35)
High-density lipoprotein [Mean (Standard Deviation); unit: mg/dL] | 41 (12) | 43 (10) | 48 (18) | 44 (22) | 44 (16)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 121 (74) | 111 (57) | 112 (51) | 153 (145) | 123 (88)
systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 136 (22) | 140 (16) | 135 (20) | 142 (21) | 138 (20)
diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 80 (16) | 81 (12) | 78 (11) | 83 (13) | 80 (13)
Weight [Mean (Standard Deviation); unit: kg] | 111 (25) | 106 (26) | 112 (21) | 113 (25) | 110 (24)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 41 (9) | 41 (9) | 42 (7) | 42 (10) | 41 (9)
Waist circumference [Mean (Standard Deviation); unit: cm] | 119 (16) | 118 (16) | 120 (14) | 115 (21) | 118 (17)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Body weight at five-month follow-up minus baseline body weight. Body weight is measured in pounds
Time Frame: five-month follow-up compared to baseline
Population: Analysis was based on those completing the five-month program and not lost to follow-up after five months.
Measure: Mean (Standard Error); unit: pounds
Arm/Group | Tele-health Home Monitoring | Self-Directed Group | TrestleTree Telephone Coaching | Home Monitoring + Telephone Coach
Number analyzed (Participants) | 35 | 31 | 33 | 27
pounds | -1.7 (1.1) | -.2 (1.9) | -4.3 (1.4) | -3.0 (1.9)
Statistical Analysis 1: Comparison: Tele-health Home Monitoring vs Self-Directed Group vs TrestleTree Telephone Coaching vs Home Monitoring + Telephone Coach; The null hypothesis is that there are no differences in the outcome across groups; Test type: Superiority; p = .296, ANOVA

2. Primary Outcome: Change in Waist Circumference
Description: Waist circumference at five-month follow-up minus waist circumference at baseline. Waist circumference is measured in centimeters.
Time Frame: five-month follow-up compared to baseline
Population: Analysis was done using those who completed the five-month programs and were not lost to follow-up at five months.
Measure: Mean (Standard Error); unit: centimeters
Arm/Group | Tele-health Home Monitoring | Self-Directed Group | TrestleTree Telephone Coaching | Home Monitoring + Telephone Coach
Number analyzed (Participants) | 35 | 31 | 33 | 27
centimeters | -.1 (.7) | -.5 (.8) | -1.5 (.9) | -.6 (1.6)
Statistical Analysis 1: Comparison: Tele-health Home Monitoring vs Self-Directed Group vs TrestleTree Telephone Coaching vs Home Monitoring + Telephone Coach; The null hypothesis is that there are no differences in the outcome across groups; Test type: Superiority; p = .787, ANOVA

3. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change is systolic blood pressure (mmHg) from baseline to five-month follow-up.
Time Frame: Systolic blood pressure (mmHg) at five months minus systolic blood pressure at baseline.
Population: Outcome results are for those who completed the study through five-months and were not lost to follow-up.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Tele-health Home Monitoring | Self-Directed Group | TrestleTree Telephone Coaching | Home Monitoring + Telephone Coach
Number analyzed (Participants) | 35 | 31 | 33 | 27
mm Hg | -4.7 (2.9) | -1.6 (2.5) | -3.4 (3.2) | -9.6 (3.6)
Statistical Analysis 1: Comparison: Tele-health Home Monitoring vs Self-Directed Group vs TrestleTree Telephone Coaching vs Home Monitoring + Telephone Coach; The null hypothesis is that there are no differences in the outcome across groups; Test type: Superiority; p = .340, ANOVA

4. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change in diastolic blood pressure (mmHg) from baseline to follow-up.
Time Frame: Diastolic blood pressure (mmHg) at five months minus diastolic blood pressure at baseline.
Population: Analysis is based on those who completed the study through five months and were not lost to follow-up.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Tele-health Home Monitoring | Self-Directed Group | TrestleTree Telephone Coaching | Home Monitoring + Telephone Coach
Number analyzed (Participants) | 35 | 31 | 33 | 27
mm Hg | -2.5 (1.9) | -1.3 (1.6) | -1.6 (2.0) | -5.3 (2.2)
Statistical Analysis 1: Comparison: Tele-health Home Monitoring vs Self-Directed Group vs TrestleTree Telephone Coaching vs Home Monitoring + Telephone Coach; The null hypothesis is that there are no differences in the outcome across groups; Test type: Superiority; p = .502, ANOVA

5. Secondary Outcome: Change in HbA1c
Description: Change in HbA1c value from baseline to five-month follow-up among those completing the study through five months.
Time Frame: five months
Population: The analysis was based on those who completed the study through five months and who had both baseline and follow-up lab results available from the electronic medical record.
Measure: Mean (Standard Error); unit: change in HbA1c percentage
Arm/Group | Tele-health Home Monitoring | Self-Directed Group | TrestleTree Telephone Coaching | Home Monitoring + Telephone Coach
Number analyzed (Participants) | 18 | 14 | 14 | 7
change in HbA1c percentage | -.01 (.21) | .19 (.13) | .11 (.19) | -.01 (.08)
Statistical Analysis 1: Comparison: Tele-health Home Monitoring vs Self-Directed Group vs TrestleTree Telephone Coaching vs Home Monitoring + Telephone Coach; The null hypothesis is that the outcome does not differ across the four groups; Test type: Superiority; p = .860, ANOVA

6. Secondary Outcome: Change in Triglycerides
Description: Change from baseline to five month follow-up in triglyceride level.
Time Frame: five months
Population: The analysis was based on those subjects completing the study through five months and for whom triglyceride levels were available in the study sites' electronic medical records.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Tele-health Home Monitoring | Self-Directed Group | TrestleTree Telephone Coaching | Home Monitoring + Telephone Coach
Number analyzed (Participants) | 16 | 14 | 8 | 11
mg/dL | -5.3 (8.9) | 3.8 (7.2) | 12 (9.2) | 2 (10.1)
Statistical Analysis 1: Comparison: Tele-health Home Monitoring vs Self-Directed Group vs TrestleTree Telephone Coaching vs Home Monitoring + Telephone Coach; The null hypothesis is that the outcome does not differ across the four groups; Test type: Superiority; p = .634, ANOVA

7. Secondary Outcome: Change in Total Cholesterol
Description: Change in total cholesterol level from baseline to five-month follow-up.
Time Frame: five months
Population: The analysis is based on subjects completing the study through five months and who had total cholesterol lab values available in the study sites' electronic medical records.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Tele-health Home Monitoring | Self-Directed Group | TrestleTree Telephone Coaching | Home Monitoring + Telephone Coach
Number analyzed (Participants) | 16 | 14 | 8 | 11
mg/dL | -10.1 (9.1) | -6.1 (4.8) | -.8 (11.0) | -6.9 (4.7)
Statistical Analysis 1: Comparison: Tele-health Home Monitoring vs Self-Directed Group vs TrestleTree Telephone Coaching vs Home Monitoring + Telephone Coach; The null hypothesis is that there is no difference in the outcome across the four treatment groups; Test type: Superiority; p = .879, ANOVA

8. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change from baseline to five-month follow-up in fasting plasma glucose level.
Time Frame: five months
Population: The analysis is based on those subjects who completed the study through five months and who had fast plasma glucose lab values available in the study sites' electronic medical record.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Tele-health Home Monitoring | Self-Directed Group | TrestleTree Telephone Coaching | Home Monitoring + Telephone Coach
Number analyzed (Participants) | 19 | 16 | 14 | 14
mg/dL | 13.6 (9.8) | 4.1 (5.9) | 5.9 (20.1) | 10.9 (9.4)

ADVERSE EVENTS:
Time Frame: Five months from baseline (randomization) through five-month follow-up
Description: The adverse event data summary includes all adverse events identified for the initially randomized 202 subjects, not just for the 126 subjects who completed the study. That is because adverse events identified over the course of the five-month study include identified adverse events for those who subsequently did not complete the study. For example, a subject may have had an adverse event in the second month but have been lost to follow-up by the end of month five when the study ended.
Arm/Group | Tele-health Home Monitoring | Self-Directed Group | TrestleTree Telephone Coaching | Home Monitoring + Telephone Coach
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/51 | 0/52 | 0/49
Serious Adverse Events (participants affected / at risk) | 14/50 | 20/51 | 22/52 | 19/49
Other Adverse Events (participants affected / at risk) | 1/50 | 3/51 | 6/52 | 3/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tele-health Home Monitoring (N=50) | Self-Directed Group (N=51) | TrestleTree Telephone Coaching (N=52) | Home Monitoring + Telephone Coach (N=49)
Hospitalization and/or emergency department visit (Surgical and medical procedures) | 14 (20) | 18 (29) | 19 (31) | 19 (27) — Hospitalization for any reason or an emergency department visit for any reason
unexpected outpatient clinic visit (General disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1) — Unexpected/unplanned outpatient clinic visits for emergent conditions.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tele-health Home Monitoring (N=50) | Self-Directed Group (N=51) | TrestleTree Telephone Coaching (N=52) | Home Monitoring + Telephone Coach (N=49)
mild or moderate unanticipated health events (General disorders) | 1 (1) | 3 (3) | 6 (6) | 3 (3) — Includes (1) unanticipated outpatient clinic visits and (2) significant changes in reported health status not resulting in emergency department visits or hospitalization and deemed unrelated or unlikely to be related to the study interventions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No